CLINICAL TRIAL: NCT04186702
Title: New Concepts in Diabetic Macular Edema (DME) Ranibizumab and Focal/Direct Laser for Chronic Diabetic Macular Edema With Vision Impairment
Brief Title: New Concepts in Diabetic Macular Edema (DME)
Acronym: DME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, khaled hamdi elbaklish, principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FWA000017585 FMASU22/2017
Record Dates: First submitted 2019-11-30; First posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, With Complications
Keywords: macula-injection- laser- ranibizumab-edema-thickness
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Intervention Model Description: interventional model
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A clinical trial design strategy in which parties involved in the trial, the investigator and participants, do not know which participants have been assigned which interventions. Type of masking include: double-blind masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- visual acuity letter score (Active Comparator): visual acuity letter score is used to compare between the two groups after interventional procedures
  Interventions: Procedure: INTRAVITREAL RANIBIZUMAB INJECTION
- macular thickness(CST) (Active Comparator): macular thickness(CST)is used to compare between the two groups after interventional procedures
  Interventions: Procedure: INTRAVITREAL RANIBIZUMAB INJECTION

INTERVENTIONS:
Procedure: INTRAVITREAL RANIBIZUMAB INJECTION — interventions involving RANIBIZUMAB INJECTION 0.5 mg (0.05 mL of 10 mg/mL solution)
  Other Names: focal/direct argon laser

SUMMARY:
Intravitreal ranibizumab injection procedure is simple and effective. In management of chronic DME there is no clear anatomical endpoint. Visual stability is the primary aim. Argon focal laser therapy can be the safe second choice. The combined therapy is successful and practical for chronic DME patients.

DETAILED DESCRIPTION:
Settings and Design: Randomized clinical study

Subjects and Methods:

investigators randomly assigned 150 adults (the average age was 59.32 years ±2.79) with chronic diabetic macular edema involving the macular center for repeated ranibizumab injections (group A-75) or focal/direct argon laser after repeated ranibizumab injections (group B-75). The outcomes were the changes in visual acuity letter score and the central subfield thickness (CST) from baseline to one year. visual-acuity Letter score, and CST were analyzed with independent t-test and Mann Whitney-test. General linear model with multivariate analysis was used for visual acuity letter score, and CST in both groups.

ELIGIBILITY:
Inclusion Criteria:

* focal maculopathy
* diffuse macular edema
* diffuse macular edema with ischemic changes

Exclusion Criteria:

* ischemic maculopathy that was associated with grades of non-proliferative changes, or capillary drop out zones presented in the periphery of the macula
* patients with history of stroke or transient ischemic attack
* hypersensitivity to ranibizumab or any component of the ranibizumab formulation
* uncontrolled glaucoma in either eye (intraocular pressure [IOP] >24 mmHg with medication)
* evidence of vitreomacular traction (in either eye)
* active proliferative diabetic retinopathy (study eye)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2016-10-01 (Actual); Study Completion 2017-09-09 (Actual)

PRIMARY OUTCOMES:
visual acuity letter score | one-year follow up
  The visual acuity letter score at one-year
central subfield thickness (CST) | one-year follow up
  the mean CST observed at one-year

SECONDARY OUTCOMES:
patient compliant-complications | one-year follow up
  subjective symptoms

IPD SHARING:
Plan to Share IPD: No
Data processed and saved in eye center in the college